CLINICAL TRIAL: NCT05424601
Title: Testing the Modular Intervention in a Small-scale Study of Game Based Cognitive Change ER Skills Coaching with or Without EMI
Brief Title: Intervention in a Small-scale Study of Game Based Cognitive Change Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D of Clinical Psychology, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RETthinkEMOTIONS3
Record Dates: First submitted 2022-06-15; First posted 2022-06-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Emotion Regulation
Keywords: online therapeutic game; emotional problems; emotional regulation; children and adolescents
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rethink game plus PsyPills (Experimental): Rethink game followed by PsyPills
  Interventions: Behavioral: Rethink game; Behavioral: PsyPills
- Rethink Game (Experimental): Rethink game only
  Interventions: Behavioral: Rethink game
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Rethink game — REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention to reduce emotional symptoms of children and adolescents.
  Arms: Rethink Game; Rethink game plus PsyPills
Behavioral: PsyPills — PsyPills is a mobile app designed to provide personalized psychological pills
  Arms: Rethink game plus PsyPills

SUMMARY:
This activity will have the objectives of preliminary testing user satisfaction, the feasibility of the platform and its preliminary efficacy

DETAILED DESCRIPTION:
Preliminary efficacy will be tested in an emotion-regulation framework. Children included in this study will be allocated to play Level 4 of the REThink game on cognitive change or to no intervention Control condition. Children and adolescents in the intervention group will be distributed afterwards in two groups: with or without ecological momentary intervention (EMI) using the PsyPills app for following-up with the cognitive change ER personalized strategy reminder during a real exam situation. Outcomes considered will be stress reactivity (both subjective and physiological) using EMA before, during and after the test (Colombo et al., 2020), and cognitive change, namely irrational and rational beliefs, and reflective functioning improvements.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents between 10 and 16 years old
* provided written parental consent
* able to access mobile/internet applications on their device

Exclusion Criteria:

* Intellectual disability or physical limitations precluded the use of the computer program
* Had a major mental health disorder

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 165 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Levels of rational and irrational beliefs | Baseline
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Changes in levels of rational and irrational beliefs | Post-intervention (one week after the intervention)
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Emotion regulation abilities | Baseline
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.
Changes in emotion regulation abilities | Post-intervention (one week after the intervention)
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.

CONTACTS AND LOCATIONS:
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No